CLINICAL TRIAL: NCT05680493
Title: Comparison of Dry Needling and Manual Pressure Release for Managing Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/20
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling; Diathermy

STUDY DESIGN:
Intervention Model Description: randomized control trial which will consist of two groups, control and experimental
Who Masked: Participant
Masking Description: participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Total 12 sessions of trigger point dry needling at lumbar muscles with Hot pack,with 3 sessions per week
  Interventions: Procedure: Dry needling; Procedure: Heat therapy
- manual pressure release (Active Comparator): Hot pack for 15 min then manual pressure release
  Interventions: Procedure: Manual pressure release; Procedure: Heat therapy

INTERVENTIONS:
Procedure: Manual pressure release — lengthens the muscle up to the increasing resistance, then gradually applies gentle pressure on MTrp until fingers feels a definite increase in tissue resistance (first barrier). Pressure would maintain until clinician sense relief of tension
  Arms: manual pressure release
Procedure: Dry needling — A filiform needle is inserted at 45 degree in to trigger point and then twirl the needle up and down to release trigger point
  Arms: Dry needling
Procedure: Heat therapy — Hydro collator pack will be placed on affected area for relaxation and pain relief for 15 min

SUMMARY:
This study will compare the effect of dry needling and manual pressure in patients having low back pain in terms of pain and disability. There will be two groups ; experimental and control. Half of study group will receive dry needling session along with hot pack. Half of study group will receive manual pressure technique along with hot pack.

DETAILED DESCRIPTION:
The study is Randomized Control Trail , which is being conducted in fauji foundation hospital and Foundation University College Of Rehabilitation (oct 2022-feb 2023) . Sample size of 50 individual was calculated using epitool with 95% confidence interval (CI), and power 80%. sample will be collected through pilot study .

both groups will recieve conventional physiotherapy protocol (hot pack) Assessment will be done on baseline, and 4th week .

ELIGIBILITY:
Inclusion Criteria:-

* age between 30-60
* pateint with subacute and chronic low back pain at least last 6 months.
* pateint with active MTrps.

Exclusion Criteria:

* patient with fibromyalgia
* pregnant females
* patient with chronic diseases (osteoporosis, lungs disease and diabetes)
* patient with musculoskeletal injuries
* patient that are using any medication to relief pain like analgesic or muscle relaxants
* Any treatment for back pain in same period of research.
* patient having any radiculopathies or discogenic low back pain

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 4 weeks
  visual analogue scale
functional disability | 4 weeks
  functional disability will be measured through oswestry disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan